CLINICAL TRIAL: NCT05877248
Title: The Knowledge and Practice of Preoperative Clear Liquid Diet Fasting Among Medical Staff in a Medical School Hospital.
Brief Title: Preoperative Clear Liquid Diet Fasting; Survey Among Medical School Physician
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, assistance professor, Mahidol University
Other Study IDs: SI 325/2566
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-03

CONDITIONS: Fasting Before Operation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine knowledge and practice about liquid diet fasting among physicians in a Quaternary-care academic center

study decide: questionnaire based study to ask concerning and knowledge and practice about liquid diet fasting and other diet fasting.

ELIGIBILITY:
Inclusion Criteria:

* physician who have opportunity to order fasting for surgical patient.

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: physician who have opportunity to order fasting for surgical patient.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Score of multiple-choice question test about fasting before operation in physician of medical school. | 1 year
  Multiple-choice question for access knowledge about fasting before operation in physician of medical school. Possible score range from 0 (poor knowledge) to 8 (excellence knowledge).

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of medicine Siriraj hospital, Mahidol University, Bangkok
  - faculty of medicine Siriraj hospital, Bangkok